CLINICAL TRIAL: NCT05899894
Title: Neurally Adjusted Ventilatory Assist (NAVA) Use in Infants With Acute Viral Bronchiolitis: a Randomised, Crossover Feasibility Study
Brief Title: NAVA in Infants With Acute Viral Bronchiolitis: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 217195
Record Dates: First submitted 2022-12-08; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-02

CONDITIONS: Acute Viral Bronchiolitis
MeSH Terms: interventions — Interactive Ventilatory Support

STUDY DESIGN:
Intervention Model Description: Patients will act as their own control. They will be randomised on day 1 to receive either standard dose or low dose morphine and on day two they will receive the alternate dose. Ventilation levels will be titrated as per a titration protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A - Low dose morphine (Active Comparator): Low dose morphine 5mcg/kg/hr
  Interventions: Device: Neurally Adjusted Ventilatory Assist
- B- standard dose morphine (Active Comparator): Standard dose morphine 20mcg/kg/hr
  Interventions: Device: Neurally Adjusted Ventilatory Assist

INTERVENTIONS:
Device: Neurally Adjusted Ventilatory Assist — NAVA mode will be titrated as per protocol alongside titration of PEEP levels. Peep will be titrated for all NAVA levels in a descending order 10,5,0 NAVA level will be titrated in an ascending order 0.5, 1.0, 1.5, 2.0 at each PEEP level

SUMMARY:
This exploratory intervention feasibility study aims to evaluate the use of a novel mode of ventilation known as Neurally adjusted ventilatory assist (NAVA) in infants with acute viral bronchiolitis.

The main aims are:

1. To determine whether an optimal combination of NAVA support level and Positive End Expiratory Pressure (PEEP) exists that can:

   1. maximise aspects of respiratory muscle unloading and
   2. minimize air trapping
2. To evaluate the impact of two morphine infusion doses on comfort levels and respiratory drive (standard = 20mcg/kg/hr, low = 5mcg/kg/hr) during ventilation titration.

Patients will act as their own control and will be randomly allocated to receive either standard or low dose morphine. They will receive the alternate dose on day 2. During each period of morphine dosing ventilation levels will be titrated and vital signs, respiratory parameters and comfort b scales will be recorded.

DETAILED DESCRIPTION:
This study is a Randomised, non-blinded, crossover (morphine dose), mode of ventilation feasibility study to evaluate the use of NAVA in infants with acute viral bronchiolitis.

Background and study aims:

This study aims to evaluate a novel mode of mechanical ventilation (breathing machine), Neurally Adjusted Ventilatory Assist (NAVA), in infants admitted to the paediatric intensive care unit (PICU) with acute viral bronchiolitis. This respiratory illness accounts for 12% of PICU admissions nationally. Current modes of ventilation are inefficient, often requiring prolonged use of sedative drugs for comfort and to improve ease of ventilation (synchronicity). Consequences of prolonged sedative use are muscle wastage including the respiratory muscles, increased risk of developing secondary infections and the potential for withdrawal from medication symptoms.

NAVA is a mode of ventilation that is delivered using our current ventilators (breathing machines). However, it differs from current modes by providing respiratory support in proportion to the signal from the brain to move the diaphragm, this is achieved via measurement of electrical activity of the diaphragm (the main muscle used to initiate a breath). This is measured by using a modified version of the patients' feeding tube (which is used in PICU to feed patients whilst on a ventilator).

Research in children to date has demonstrated that NAVA, compared to other ventilatory modes, allows for improved ventilator synchrony, reduced work of breathing and potentially less sedative use. This is consistent with our clinical impression (we have been using NAVA in an ad hoc way for >5 years). Although some of these studies included infants with bronchiolitis, the findings were not specific to this patient group. Of note, we do not yet know how to optimise NAVA settings in bronchiolitis, and whether current common sedative drugs (e.g. morphine) affect this, by decreasing respiratory drive excessively (potentially compromising NAVA utility).

We will evaluate how to optimise NAVA settings when compared to conventional ventilation in infants with acute viral bronchiolitis admitted to PICU. A range of NAVA settings will be systematically evaluated over two periods on consecutive days (maximum 4 hours per period per day). Observation of the effects of different levels of NAVA support on synchronicity, work of breathing and changes in physiological parameters will take place. Patients will also receive 2 different adjustments to their morphine infusions in random order on the consecutive days: standard dose morphine (20mcg/kg/hr) and low dose morphine (5mcg/kg/hr). Both morphine doses are within the range currently used clinically. Patient comfort will be assessed frequently throughout, and the effects of morphine on diaphragmatic neural activity will be recorded.

Who can participate:

* Infants aged > 36 weeks corrected gestation and < 1 year of age
* Admitted to PICU with acute viral bronchiolitis within 48 hours of admission
* Likely to require mechanical ventilation for > 24 hours after enrolment
* Able to pass a nasogastric tube

What does the study involve:

Within 48 hours parents/carers of patients admitted with a primary diagnosis of acute viral bronchiolitis who meet the inclusion criteria will be approached by a member of the direct healthcare team and invited to take part in the study. The pre-existing feeding tubes will be replaced with NAVA catheters by the bedside nurse or research team. Ventilation modes will be titrated on 2 consecutive days accompanied by two different Morphine doses delivered to the participant in random order. Participants will be randomised to receive either standard dose morphine (20mcg/kg/hr) or low dose morphine (5 mcg/kg/hr). These doses have been chosen to reflect current clinical practice and also using knowledge of morphine kinetics/dynamics on infant respiratory drive.

Ventilation titration involves changes in NAVA level which increase over time and changes in PEEP which decrease over time to assess the ventilator setting that the patient responds to in terms of the outcome measures. This will enable identification of the optimum ventilation strategy for that participant. Titration will occur over time on 2 consecutive days as outlined above. There will be a wash in period of 5-10 minutes for each change in ventilator setting and a period of 5 minutes when the recordings of the outcome measures will take place.

Baseline recordings will be taken for current ventilator settings, vital signs and respiratory measures and COMFORT-behavioral scale (comfort/pain scale). Study procedures will be timed to accommodate routine care such as daily physiotherapy sessions.

Benefits and risks:

Due to changes in ventilation settings during the two NAVA/PEEP titration periods (one per day) there is the potential for the child to experience changes in their comfort levels and/or physiological parameters. These will be continuously monitored by the researchers and the clinical bedside team. If the patient experiences discomfort during the study period as expressed by a COMFORT-b the patient will be returned to the previous ventilator settings and the reasons for discomfort will be assessed. Pain and sedation guidance will be adhered to as per usual care.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged > 36 weeks corrected gestation and < 1 year of age
* Admitted to PICU with acute viral bronchiolitis within 48 hours of admission
* Likely to require mechanical ventilation for > 24 hours after enrolment
* Able to pass a nasogastric tube

Exclusion Criteria:

* Apnoea as a primary reason for ventilation in the absence of respiratory symptoms
* History of gastro-intestinal bleeds in previous 30 days or significant coagulopathy
* Facial trauma or surgery
* Known neuro-muscular disease or diaphragmatic palsy
* Haemodynamic instability (requiring inotropes)

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Changes to neuroventilatory efficiency when ventilation parameters are titrated | Measures will be recorded during the intervention
  Measured by a change in neuro-ventilatory efficiency (NVE) during titration of ventilation settings
  NVE is measured as a ratio between electrical activity of the diaphragm (Edi) and patient's tidal volume during inspiration (Edi/Tv). An improvement in NVE can be demonstrated by a decrease in Edi without a fall in Tv.
Changes to neuromuscular efficiency when ventilation parameters are titrated. | Measures will be recorded during the intervention
  Measured by a change neuro-muscular efficiency (NME) during changes in ventilation settings
  NME measures Edi against the generated airway pressure during an occlusion (P0.1) thus providing an estimate of inspiratory driving pressure normalized to inspiratory neural inspiratory effort. This will be presented as a ratio: Paw (airway pressure) - PEEP)/ Edi.
Changes to air trapping when ventilation parameters are titrated | Measures will be recorded immediately after each intervention
  A forced deflation (FD) will require pressure to be applied to the thoracic area to mimic a forced exhalation - pressure loops will be recorded via the servo-i during this time. This will give an idea of forced vital capacity and the amount of airway resistance as FD causes dynamic compression of the airways. Residual volume will indicate level of air-trapping occurring.
  Forced Expiratory Volume (FEV) will be measured at the end of each PEEP level to assess the residual volume, a marker of air-trapping to assess whether PEEP titration overcomes intrinsic PEEP. This will be measured using a standardised physiotherapy technique. A large inflation breath (approx. 40cmH20) will be administered to the patient and held for 3 seconds followed by a manual compression, the ventilator will record flow loops from this compression - the degree of scalloping will be quantified in measuring the degree of air trapping using a validated calculation.
Change in Electrical activity of the diaphragm (Edi) when ventilator parameters are titrated | Measures will be recorded immediately after each intervention
  Edi is a reflection of the electrical activity on the diaphragm. Normal Edi is 5-15 microvolts. There would be an expectation that this would change if the ventilation is meeting the patients ventilatory demands
Maintenance of patient comfort | Measures will be recorded immediately after each intervention
  Patient comfort will be measured using a COMFORT-Behavioral Scale (COMFORT-b). The COMFORT-b scale is an observational scale that has been validated for assessing comfort in children in PICU. Pain in children from 0-3 years of age and sedation in the 0-16 year old child. A score of 0-40 with a score greater than 22 indicating discomfort.
Changes in blood pressure | Measures will be recorded immediately after each intervention
  Changes to blood pressure will be recorded to ensure they are within normal range for the child's age.
Changes in heart rate | Measures will be recorded immediately after each intervention
  Changes to heart rate heart Rate recorded to ensure they are within normal range for the child's age.
changes in respiratory rate | Measures will be recorded immediately after each intervention
  Changes in respiratory rate will be recorded to ensure they are within normal range for the child's age.
Stabilisation of vital signs | Measures will be recorded immediately after each intervention
  Changes in transcutaneous carbon dioxide (TCO2) will be recorded to ensure they are within normal range for the child's age.

SECONDARY OUTCOMES:
To assess recruitment rate | On study completion up to 1 year
  Record recruitment rates of participants
To assess retention rates | On study completion up to 1 year
  Record retention rates of participants
To assess time to recruit participants | On study completion up to 1 year
  Record how long from admission it took to consent a participant into the study
To record the incidence of adverse events | On study completion up to 1 year
  Recording of events as per Good Clinical Practice
To assess the willingness of clinicians to recruit participants | On study completion up to 1 year
  Number approached and consented per clinician

CONTACTS AND LOCATIONS:
Overall Officials: Shane Tibby, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The plan is not to share the raw data due to the exploratory nature of the study and the size of the individual data sets.